CLINICAL TRIAL: NCT01814384
Title: Medico-economic Study of Patient Matched Cutting Blocks (Ancillary) MyKnee ® LBS During Knee Arthroplasty GMK ®. Multicentric, Prospective, Controlled, Opened, Randomised Study About Medical Device.
Brief Title: Medico-economic Study of Patient Matched Cutting Blocks (Ancillary) MyKnee ® LBS During Knee Arthroplasty GMK ®.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC 12_0100
Record Dates: First submitted 2013-03-11; First posted 2013-03-19 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
Keywords: Ancillary tailored; medico-economic study,; total knee replacement; primary or secondary osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Control group will be constituted of patients with the prosthesis GMK ® without the ancillary MyKnee ® LBS.
  Interventions: Device: prosthesis GMK ® without the ancillary MyKnee ® LBS
- Matched patient (Other): Treated group will consist of patients which the GMK ® prosthesis with ancillary ® MyKnee LBS.
  Interventions: Device: Matched patient cutting blocks MyKnee ® LBS

INTERVENTIONS:
Device: prosthesis GMK ® without the ancillary MyKnee ® LBS
  Arms: Control group
Device: Matched patient cutting blocks MyKnee ® LBS
  Arms: Matched patient

SUMMARY:
Total knee arthroplasty represents over 70 000 surgical procedures per year in France, increasing about 10% each year since the early 1990s. Clinical experience shows a strong rate of success on pain relieve and improvement of knee articular function for these patients.

Longevity of the implants had been proved to depend on the biomechanical design and implantation techniques, particularly the bone cuts during the surgery. To improve the precision of these cuts, the patient matched cutting blocks developed by Medacta company allows to adapt bone cuts to the patient anatomy improving the reliability of these procedure. A reduction of surgical time and bleeding would be another benefit expected with this type of ancillary. The objective of this study is to demonstrate the advantage of patient matched cutting blocks for total knee arthroplasty on realiability for both clinical and radiological criteria, morbidity reduction during and after the procedure and also a benefit on an economic point of view.

ELIGIBILITY:
Inclusion Criteria:

all patients requiring a total knee arthroplasty line: primary or secondary osteoarthritis advanced beyond medical treatment.

Exclusion Criteria:

distorded axes or laxity requiring the establishment of constrained prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
compare the functionality of the knee after installation of a total knee replacement between the 2 groups | 2 years after
  The evaluation will use a specific score for total knee arthroplasty: Part of the Knee Society function score (KSS) measured at 1 year after surgery.

SECONDARY OUTCOMES:
to assess knee function by autoquestionnaire KOOS, the KSS knee score, operative time, procedure bleeding, reliability of the ancillary | 2 years after
medico-economic evaluation type "Cost minimization" | 2 years after
  * Compare the costs of implementing the two strategies (A and B) taking into account the resources consumed (operative time, anesthetic drugs, blood bags ...).
  * Determine the least costly therapeutic intervention and medico-economic impact in the current system of financing of hospital expenditure.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nantes, Nantes, France, France